CLINICAL TRIAL: NCT00871039
Title: Randomized Clinical Trial Comparing Propofol and Midazolam in Mechanically Ventilated Critically Ill Patients With Alcohol Use Disorders: An Open Label Pilot Study
Brief Title: Pilot Study Evaluating Stress Response and Immune Function in Mechanically Ventilated Patients With Alcohol Use Disorders Treated With Propofol or Midazolam
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to logistical purposes
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VCU IRB HM12035
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Alcoholism; Respiration, Artificial
Keywords: Alcoholism; Mechanical ventilation
MeSH Terms: conditions — Alcoholism; Respiratory Aspiration | interventions — Propofol; Midazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Experimental): Patients to be sedated for up to 72 hours with study drug propofol
  Interventions: Drug: Propofol
- Midazolam (Experimental): Patients to be sedated for up to 72 hours with study drug midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Propofol — Patients to be sedated for up to 72 hours with study drug propofol
  Arms: Propofol
Drug: Midazolam — Patients to be sedated for up to 72 hours with study drug midazolam
  Arms: Midazolam

SUMMARY:
The aim of this study is to evaluate the effects of the sedatives propofol and midazolam on stress response and immune function in critically ill patients with alcohol use disorders who are undergoing mechanical ventilation.

DETAILED DESCRIPTION:
No detailed description

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcohol use disorders
* Need for invasive mechanical ventilation
* Need for continuous intravenous infusion of sedative(s)

Exclusion Criteria:

* Age < 18 years
* Pregnant women
* Prisoners
* Receiving propofol prior to randomization
* Patient experiencing active alcohol withdrawal
* Immunosuppression
* Shock
* Attending physician does not feel patient is candidate to receive either propofol or midazolam
* Patient has contraindication(s) to receiving either propofol or midazolam
* Inability to enroll patient within 96 hours after initiation of mechanical ventilation
* Transfer from another intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Stress response and immune function. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Wit, M.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Virginia Commonwealth University Medical Center (formerly known as Medical College of Virginia), Richmond, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No